CLINICAL TRIAL: NCT05256043
Title: Case-control Investigation of Critically Ill Patients With Newly Diagnosed Diabetes: Clinical Characteristics, Glucose Metrics and Outcomes
Brief Title: Investigation of Critically Ill Patients With Newly Diagnosed Diabetes
Status: Completed | Type: Observational
Sponsor: Stamford Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TSH_InternalMedicine_2021010
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Glucose Metrics; Outcome Evaluation; Intensive Care Unit
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Target Population: Adult patients age ≥ 18 admitted to the Stamford Hospital ICU between 9/14/11 and 11/30/19 with HbA1c available on admission and at least 4 blood glucose (BG) tests during ICU stay. Two groups were created; patients with previously undiagnosed diabetes (NDDM) compared to those with known diabetes (KDM) at the time of admission to the intensive care unit (ICU).
  Interventions: Diagnostic Test: Diabetes Diagnosis

INTERVENTIONS:
Diagnostic Test: Diabetes Diagnosis — HbA1c > 6.5%

SUMMARY:
The purpose of this study is to investigate the clinical outcomes and glucose control metrics of critically ill patients with previously undiagnosed diabetes compared to those with known diabetes at the time of admission to the intensive care unit (ICU).

DETAILED DESCRIPTION:
This case control study compares previously undiagnosed diabetic patients (defined as HbA1c > 6.5% and no history of diabetes), to those with known diabetes, using 1:1 matching. Patients met inclusion criteria by having HbA1c available on ICU admission and at least four blood glucose tests during their ICU stay. Primary outcomes included ICU length of stay and inpatient mortality. Secondary outcomes included glucose metrics: mean blood glucose, coefficient of variation and percentage of patients who developed hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:20

* Patients admitted between 9/14/2011 and 11/30/19 with HbA1c available on admission and at least four documented blood glucose tests during their ICU stay.

Exclusion Criteria:

* Patients admitted for diabetic ketoacidosis.
* Patients admitted to the ICU following cardiovascular surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU where they were subsequently diagnosed for the first time with diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 1777 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Inpatient mortality | 2011-2019
  Estimates the risk of short-term mortality based on data from the initial 24 hours of intensive care unit (ICU) admission. Acute Physiology and Chronic Health Evaluation (APACHE) IV
Length of hospital Stay | 2011-2019
  Total days spent admitted to the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Stamford Health, Stamford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No